CLINICAL TRIAL: NCT06655246
Title: A Phase 1a/1b Study of the Safety, Pharmacokinetics, and Antitumor Activity of the Oral Menin Inhibitor Ziftomenib in Combination With Imatinib in Patients With Advanced Gastrointestinal Stromal Tumors (GIST) After Imatinib Failure
Brief Title: A Study of Ziftomenib in Combination With Imatinib in Patients With Advanced Gastrointestinal Stromal Tumors (GIST)
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Kura Oncology, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KO-MEN-015
Record Dates: First submitted 2024-10-14; First posted 2024-10-23 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Gastrointestinal Stromal Tumor (GIST); Gastrointestinal Stromal Cancer; Gastrointestinal Stromal Neoplasm; Gastrointestinal Stromal Tumor, Malignant; Gastrointestinal Stromal Cell Tumors
Keywords: Gastrointestinal Stromal Tumor; Gastrointestinal Stromal Cancer; Gastrointestinal Stromal Neoplasm
MeSH Terms: conditions — Gastrointestinal Stromal Tumors | interventions — Imatinib Mesylate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Dose Escalation (Experimental): Ziftomenib plus imatinib
  Interventions: Drug: ziftomenib; Drug: imatinib mesylate
- Recommended Phase 2 Dose Determination (Experimental): Ziftomenib plus imatinib
  Interventions: Drug: ziftomenib; Drug: imatinib mesylate
- Dose Expansion (Experimental): Ziftomenib plus imatinib
  Interventions: Drug: ziftomenib; Drug: imatinib mesylate

INTERVENTIONS:
Drug: ziftomenib — menin inhibitor
Drug: imatinib mesylate — kinase inhibitor
  Other Names: Gleevec

SUMMARY:
In this clinical trial, the safety, tolerability, and preliminary antitumor activity of ziftomenib in combination with imatinib will be evaluated in adults with gastrointestinal stromal tumors (GIST) who have been treated previously with imatinib.

ELIGIBILITY:
Key Inclusion Criteria:

* Documented diagnosis of advanced/metastatic KIT-mutant GIST.
* Documented disease progression on imatinib as current or prior therapy.
* Eastern Cooperative Oncology Group (ECOG) performance status of ≤2 at screening.
* At least 1 measurable lesion per RECIST v1.1 modified for GIST.
* Negative pregnancy test for participants of childbearing potential.
* Adequate organ function per protocol requirements.
* Resolution of all clinically significant toxicities from prior therapy to <Grade 1 (or participant baseline) within 1 week before the first dose of study intervention.
* Participant, or legally authorized representative, must be able to understand and provide written informed consent before the first screening procedure.

Key Exclusion Criteria:

* Diagnosis of GIST without a KIT mutation or with a T670X KIT mutation.
* History of prior or current cancer that has potential to interfere with obtaining study results.
* Received a prohibited medication, including investigational therapy, less than 14 days or within 5 drug half-lives before the first dose of study intervention.
* Active central nervous system metastases.
* Uncontrolled intercurrent illness, including, but not limited to protocol defined cardiac disease.
* Mean corrected QT interval (QTcF) greater than 470ms.
* Left ventricular ejection fraction (LVEF) <50%.
* Major surgery within 2 weeks before the first dose of study intervention.
* Is pregnant or breastfeeding.
* Gastrointestinal abnormalities that may impact taking study intervention by mouth.
* Actively bleeding, excluding hemorrhoidal or gum bleeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 157 (Estimated)
Dates: Start 2025-03-27 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Dose Escalation: Dose Limiting Toxicity (DLT) | Cycle 1 (first 28 day cycle)
  Rate of DLTs per dose level
Descriptive statistics of Adverse Events (AEs) | First dose of ziftomenib up to and including 28 days after last dose of ziftomenib, or if the participant is lost to follow-up, whichever comes first
  Per the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) v5.0
Dose Expansion: Clinical benefit rate (CBR) | Up to 2 years following start of treatment with ziftomenib
  CBR is the rate of participants achieving complete response (CR), partial response (PR), or stable disease (SD), assessed per Response Criteria in Solid Tumors (RECIST) v1.1 modified for GIST

SECONDARY OUTCOMES:
Recommended Phase 2 Dose Determination and Dose Expansion: CBR | Up to 2 years following start of treatment with ziftomenib
  CBR is CR + PR + SD assessed per RECIST v1.1 modified for GIST
Overall Response Rate (ORR) | Up to 2 years following start of treatment with ziftomenib
  ORR is CR + PR assessed per RECIST v1.1 modified for GIST
Progression Free Survival (PFS) | Up to 2 years following start of treatment with ziftomenib
  Assessed per RECIST v1.1 modified for GIST
Duration of Response (DoR) | Up to 2 years following start of treatment with ziftomenib
  Defined as the time from the first response (CR or PR assessed per RECIST v1.1 modified for GIST) to disease progression or death from any cause
Overall Survival (OS) | Up to 2 years following start of treatment with ziftomenib
  Defined as the time from first dose of ziftomenib or imatinib (whichever is dosed first) until death from any cause
Maximum plasma concentration (Cmax) | Day 1 of each cycle; each cycle is 28 days
  Cmax of ziftomenib
Time to maximum plasma concentration (Tmax) | Day 1 of each cycle; each cycle is 28 days
  Tmax of ziftomenib
Area under the concentration-time curve from time zero to the time of the last quantifiable concentration (AUC 0-last) | Day 1 of each cycle; each cycle is 28 days
  AUC 0-last of ziftomenib
Area under the concentration-time curve over a dosing interval (AUC tau) | Day 1 of each cycle; each cycle is 28 days
  AUC tau of ziftomenib
Maximum plasma concentration (Cmax) | Day 1 of each cycle; each cycle is 28 days
  Cmax of imatinib
Time to maximum plasma concentration (Tmax) | Day 1 of each cycle; each cycle is 28 days
  Tmax of imatinib
Area under the concentration-time curve from time zero to the time of the last quantifiable concentration (AUC 0-last) | Day 1 of each cycle; each cycle is 28 days
  AUC 0-last of imatinib
Area under the concentration-time curve over a dosing interval (AUC tau) | Day 1 of each cycle; each cycle is 28 days
  AUC tau of imatinib

CONTACTS AND LOCATIONS:
Locations (32):
- United States (32):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Mayo Clinic Cancer Center, Phoenix, Arizona
  - University of California, San Diego, La Jolla, California
  - University of Southern California, Los Angeles, California
  - University Of California, Irvine, Orange, California
  - Stanford Cancer Institute, Palo Alto, California
  - UCLA Santa Monica Medical Center, Santa Monica, California
  - University of Colorado Cancer Center, Aurora, Colorado
  - Sarah Cannon Research Institute, Denver, Colorado
  - Yale University School of Medicine, New Haven, Connecticut
  - Mayo Clinic Cancer Center, Jacksonville, Florida
  - University of Miami, Miami, Florida
  - Northwestern University, Chicago, Illinois
  - University of Iowa, Iowa City, Iowa
  - Johns Hopkins University, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Harvard University, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - Ohio State University, Columbus, Ohio
  - Oregon Health & Science University, Portland, Oregon
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Temple University Health System, Philadelphia, Pennsylvania
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Sarah Cannon Research Institute, Dallas, Texas
  - University of Texas, Houston, Texas
  - University of Texas Health Science Center, San Antonio, Texas
  - University of Utah, Salt Lake City, Utah
  - Medical College of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No